CLINICAL TRIAL: NCT06448962
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Trial to Evaluate the Efficacy and Safety of Co-administrated AD-2021 and AD-2022 in Patients With Primary Hypercholesterolemia and Essential Hypertension
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of Co-administrated AD-2021 and AD-2022
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-202P3
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Hypertension, Essential; Primary Hypercholesterolemia
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): AD-2021, AD-2022
  Interventions: Drug: AD-2021; Drug: AD-2022
- Active Comparator 1 (Active Comparator): AD-2021, AD-2022 placebo
  Interventions: Drug: AD-2021; Drug: AD-2022 Placebo
- Active Comparator 2 (Active Comparator): AD-2022, AD-2021 placebo
  Interventions: Drug: AD-2022; Drug: AD-2021 Placebo

INTERVENTIONS:
Drug: AD-2021 — PO, Once daily(QD), 8weeks
  Arms: Active Comparator 1; Experimental 1
Drug: AD-2022 — PO, Once daily(QD), 8weeks
  Arms: Active Comparator 2; Experimental 1
Drug: AD-2021 Placebo — PO, Once daily(QD), 8weeks
  Arms: Active Comparator 2
Drug: AD-2022 Placebo — PO, Once daily(QD), 8weeks
  Arms: Active Comparator 1

SUMMARY:
The purpose of this study is to Evaluate the Efficacy and Safety of Co-administrated AD-2021 and AD-2022

DETAILED DESCRIPTION:
Condition or disease : Primary Hypercholesterolemia and Essential Hypertension Intervention/treatment Drug : AD-2021 Drug : AD-2022 Drug : AD-2021 Placebo Drug : AD-2022 Placebo Phase : Phase 3

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects with hypertension and hyperlipidemia

Exclusion Criteria:

* Patient with known or suspected secondary hypertension
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) | Baseline, Week 8
  LDL-C change at Week 8 compared AD-2021 + AD-2022 with AD-2022
Mean sitting systolic blood pressure (MSSBP) | Baseline, Week 8
  MSSBP change at Week 8 compared AD-2021 + AD-2022 with AD-2021

CONTACTS AND LOCATIONS:
Overall Officials: Seok Min Kang, M.D., Ph.D, Principal Investigator — Yonsei Cardiovascular Hospital
Locations (1):
- Yonsei Cardiovascular Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No